CLINICAL TRIAL: NCT05029245
Title: The 8-week, Prospective, Randomized Controlled of IntraDermal Administration of Comirnaty® 6 Microgram Versus Intramuscular Comirnaty® 30 Microgram by 28 Days Interval Efficacy Study in Healthy Volunteer
Brief Title: IntraDermal Versus Intramuscular Comirnaty® Efficacy Study
Acronym: PRIDE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No financial budget support
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Department of Medical services (Unknown)
Responsible Party: Principal Investigator, Dr Subsai Kongsaengdao, Associate Professor Subsai Kongsaengdao, M.D., Department of Medical Services Ministry of Public Health of Thailand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY NO. A-03-2021
Record Dates: First submitted 2021-08-20; First posted 2021-08-31 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Covid19 Vaccine; Covid19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: The 8-week, Prospective, Randomized controlled of IntraDermal administration of Comirnaty® 6 microgram compare to Intramuscular Comirnaty® 30 microgram by 28 days interval Efficacy Study in healthy volunteers.
  There were flexible 8 arms recruitment up to type of immunological background of 1000 volunteers and availability of BNT162b2 vaccine ( initially estimated 125 volunteers. Per arm)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Sinovac 2 dosage followed by Comirnaty® 6 microgram Intradermal (Experimental): Patients who had history of Coronavac vaccine 2 dosage at least 1 month before enrollment will received Intradermal Comirnaty® vaccine 6 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®
- Sinovac 2 dosage followed by Comirnaty® 30 microgram Intramuscular (Active Comparator): Patients who had history of Coronavac vaccine 2 dosage at least 1 month before enrollment will received Intramuscular Comirnaty® vaccine 30 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®
- Aztrazeneca 1 dosage followed by Comirnaty® 6 microgram Intradermal (Experimental): Patients who had history of ChAdOX1 Cov-19 vaccine 1 dosage at least 1 month before enrollment will received Intradermal Comirnaty® vaccine 6 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®
- Aztrazeneca 1 dosage followed by Comirnaty® 30 microgram Intramuscular (Active Comparator): Patients who had history of ChAdOX1 Cov-19 vaccine 1 dosage at least 1 month before enrollment will received intramuscular Comirnaty® vaccine 30 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®
- Naive vaccine followed by Comirnaty® 6 microgram Intradermal (Experimental): Patients who had no history SAR-CoV vaccine before enrollment will received intradermal Comirnaty® vaccine 6 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®
- Naive vaccine followed by Comirnaty® 30 microgram Intramuscular (Active Comparator): Patients who had no history SAR-CoV vaccine before enrollment will received intramuscular Comirnaty® vaccine 30 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®
- Any history of vaccination with Anti-RBD< 650AU/ml followed by Comirnaty® 6 microgram Intradermal (Experimental): Patients who had history of any SAR-CoV vaccine at least 1 month before enrollment will received intradermal Comirnaty® vaccine 6 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®
- Any history of vaccination with Anti-RBD <650AU/ml followed by Comirnaty® 30 microgram Intramuscular (Active Comparator): Patients who had history of any SAR-CoV vaccine at least 1 month before enrollment will received intramuscular Comirnaty® vaccine 30 microgram 2 dosage by 28 days interval
  Interventions: Biological: Comirnaty®

INTERVENTIONS:
Biological: Comirnaty® — intradermal injection or intramuscular injection

SUMMARY:
The 8-week, Prospective, Randomized controlled of IntraDermal administration of Comirnaty® 6 microgram compare to Intramuscular Comirnaty® 30 microgram by 28 days interval Efficacy Study in 4 groups of healthy volunteer ( 1 people who complete sinovac vaccination 2 people who received 1 dosage of AstraZeneca vaccine 3 naive vaccination 4 any other vaccination not in 1-3 with anti Spike antibody less than 650 AU/ ml) . Comparison of antibody level and T cell response to SAR-CoV-2 antigen in vitro after 28 day post vaccination is primary outcome and the side effect as well as infection rate in 8 weeks is secondary outcomes.

DETAILED DESCRIPTION:
The 8-week, Prospective, Randomized controlled of IntraDermal administration of Comirnaty® 6 microgram compare to Intramuscular Comirnaty® 30 microgram by 28 days interval Efficacy Study in healthy volunteer.To compare the AntiSpike antibody, ( Anti RBD ) neutralized antibody ( if possible) of SAR-CoV-2 and T-cell response after injection with Intradermal Comirnaty® 6 microgram versus Intramuscular Comirnaty® 30 microgram by 28 days interval in healthy volunteer in various immunological background groups.1000 patients with or with out vaccinated and with our without history of previous COVID-19 infection (in various immunological background ) will be recruited and received Comirnaty® 6 microgram versus Intramuscular Comirnaty® 30 microgram by 28 days interval

Inclusion Criteria:

1. Signed informed consent by any patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representatives prior to initiation of any study procedures.
2. Men and women, ≥18 years of age at time of enrollment.
3. Able to follow up the vaccination schedule.

Exclusion Criteria:

1. Patient with known hypersensitivity or intolerance to Comirnaty® or Polyethylene glycol (PEG).
2. Patient with previous receiveing mRNA vaccine ( Pfizer, Moderna or other).
3. Pregnancy with gestational age less than 12 weeks.
4. Patient with History of immunosuppessive drug ( oral , IV, IM ) of which discontinue less than 6 month or any immunological abnormality which impact to Antibody production and T cell function ( eg hypergammaglobulinemia, active immne deficiency).
5. Patient with previous used of Intravenous immunoglobulin in previous 6 month
6. Patient with history of abnormal coagulation or contraindication for intramuscular injection or intradermal injection.
7. Patient with end stage disease or disease with life expectancy less than 2 years
8. Patient with previous use of medication interfere with serum interferon other cytokine system or disease with cytokine abnormalities.
9. Patient with history of abnormal platelet or platelet dysfunction, blood coagulopathy abnormality.
10. Patient with active pulmonary tuberculosis or systemic tuberculosis, atypical non mycobacterium tuberculosis.

Primary efficacy: To compare the AntiSpike antibody, ( Anti RBD ) neutralized antibody ( if possible) of SAR-CoV-2 and T-cell response after injection with Intradermal Comirnaty® 6 microgram versus Intramuscular Comirnaty® 30 microgram by 28 days interval in healthy volunteer in various immunological background groups.

Secondary efficacy: Comparesion of infection rate in each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by any patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representatives prior to initiation of any study procedures.
2. Men and women, ≥18 years of age at time of enrollment.
3. Able to follow up the vaccination schedule.

Exclusion Criteria:

1. Patient with known hypersensitivity or intolerance to Comirnaty® or Polyethylene glycol (PEG).
2. Patient with previous receiveing mRNA vaccine ( Pfizer, Moderna or other).
3. Pregnancy with gestational age less than 12 weeks.
4. Patient with History of immunosuppessive drug ( oral , IV, IM ) of which discontinue less than 6 month or any immunological abnormality which impact to Antibody production and T cell function ( eg hypergammaglobulinemia, active immne deficiency).
5. Patient with previous used of Intravenous immunoglobulin in previous 6 month
6. Patient with history of abnormal coagulation or contraindication for intramuscular injection or intradermal injection.
7. Patient with end stage disease or disease with life expectancy less than 2 years
8. Patient with previous use of medication interfere with serum interferon other cytokine system or disease with cytokine abnormalities.
9. Patient with history of abnormal platelet or platelet dysfunction, blood coagulopathy abnormality.
10. Patient with active pulmonary tuberculosis or systemic tuberculosis, atypical non mycobacterium tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-31 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Level of Anti RBD antibody | 8 weeks
  Level of Anti RBD antibody after first and second injection
Interferon gamma level | 8 weeks
  Interferon gamma level ( production of interferon gamma Againts SAR-CoV-2 antigen in vitro after injection for 28 days

SECONDARY OUTCOMES:
COVID-19 infection | 8 weeks
  COVID-19 infection rate after first and second injection
COVID-19 death | 8 weeks
  COVID-19 death rate after first and second injection
adverse event after vaccination | 8 weeks
  adverse event rate after first and second injection

IPD SHARING:
Plan to Share IPD: No